CLINICAL TRIAL: NCT02565810
Title: An Open-labelled, Single-arm, Multicentre Clinical Study to Evaluate the Usability and Safety of the Pre-filled Pen and Pre-filled Syringe of SB5 in Subjects With Rheumatoid Arthritis
Brief Title: An Multicentre Clinical Study to Evaluate the Usability and Safety of the Pre-filled Pen and Pre-filled Syringe of SB5 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SB5-G21-RA
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — penclomedine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB5 40mg (Experimental)
  Interventions: Drug: Adalimumab PFS and Pen

INTERVENTIONS:
Drug: Adalimumab PFS and Pen

SUMMARY:
A study comparing the use of the Pre-filled Pen and Pre-filled Syringe of SB5 in Subjects with Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female aged 18-55 years at the time of signing the informed consent form.
2. Have been diagnosed as having RA according to the revised 1987 American College of Rheumatology (ACR) criteria for at least 6 months prior to Screening.
3. Subjects who are considered by the Investigator to be a suitable candidate for self-administering adalimumab treatment
4. Must be able to provide informed consent, which must be obtained prior to any study related procedures.

Exclusion Criteria:

1. Have been treated previously with any biologic agents including any tumour necrosis factor inhibitor.
2. Have a known hypersensitivity to human immunoglobulin proteins or other components of SB5.
3. Have a current diagnosis of active tuberculosis (TB), have been recently exposed to a person with active TB, or are considered to have latent TB indicated by a positive QuantiFERON® Gold test result.
4. Have had a serious infection (such as sepsis, abscess, opportunistic infections or invasive fungal infection including histoplasmosis) or have been treated with intravenous antibiotics for an infection within 8 weeks or oral antibiotics within 2 weeks prior to first dose of IP. Nonsignificant infections do not need to be considered exclusionary at the discretion of the Investigator.
5. Have a history of chronic or recurrent infection (such as chronic renal infection, chronic chest infection or recurrent urinary infection).
6. Have any of the following conditions:

   1. History of congestive heart failure (New York Heart Association Class III/IV)
   2. History of demyelinating disorders (such as multiple sclerosis or Guillain-Barré syndrome).
   3. History of any malignancy (other than lymphoproliferative disease and melanoma, see Exclusion Criteria 10.f) within the previous 5 years prior to Screening except completely excised and cured squamous carcinoma of the uterine cervix, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma.
   4. History of lymphoproliferative disease including lymphoma or melanoma.
   5. Any other disease or disorder which, in the opinion of the Investigator, will put the subject at risk if they are enrolled.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Medica Pro Familia Sp. z o.o. S.K.A. Oddzial Gdynia, Gdynia
  - Medica pro Familia Sp z o.o. S.K.A Oddzial Warszawa, Warsaw

REFERENCES:
- [Derived] Ghil J, Zielinska A, Lee Y. Usability and safety of SB5 (an adalimumab biosimilar) prefilled syringe and autoinjector in patients with rheumatoid arthritis. Curr Med Res Opin. 2019 Mar;35(3):497-502. doi: 10.1080/03007995.2018.1560211. Epub 2019 Jan 17. PMID 30561229

RESULTS

PARTICIPANT FLOW:
Groups:
- SB5 40mg: Adalimumab PFS and Pen
Period: Overall Study
Arm/Group | SB5 40mg
Started | 49
Completed | 48
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | SB5 40mg
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 167.69 (8.799)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Injection Site Pain Score Using an 11-point Visual Numeric Scale
Description: Injection site pain evaluation questionnaire will be rated on an 11-point numeric rating scale ranging from 0 (no pain) to 10 (pain as bad as it could be) at two-time points post-injection (immediately post-injection and between 15 to 30 minutes post-injection) at Weeks 0, 2, 4, and 6.
Time Frame: Difference of injection site pain score (Week 6 - Week 2)
Measure: Number (97.5% Confidence Interval); unit: Difference (scores on a scale)
Groups:
- SB5 Pen/PFS: Injection via PFS at Week 0 and Week 2 and then injection via Pen st Week 4 and then every other week thereafter up to Week 10
Arm/Group | SB5 Pen/PFS
Number analyzed (Participants) | 49
Difference (scores on a scale)
  Immediately post-injection | -0.35 [-0.99 to 0.30]
  15-30 min post-injection | -0.11 [-0.47 to 0.25]

2. Secondary Outcome: Overall Impression of SC Delivery Administration of SB5 Using Questionnaire
Description: Objective: To evaluate whether overall impressions of SC administrations at Week 2 and Week 6 were comparable between the SC administrations of SB5 via the Pen and via the PFS.
Time Frame: at Week 2 and at Week 6
Population: Only number of subjects with available assessment results at each visit were counted as 'Overall number of participants analyzed'.
Measure: Count of Participants; unit: Participants
Groups:
- Week 2 (SB5 40 mg PFS); Week 6 (SB5 40 mg Pen): 40 mg sc injection via PFS at Week 0 and Week 2 and then 40 mg sc injection via Pen st Week 4 and then every other week thereafter up to Week 10.
Arm/Group | Week 2 (SB5 40 mg PFS) | Week 6 (SB5 40 mg Pen)
Number analyzed (Participants) | 48 | 46
Participants
  Extremely Favorable | 1 | 3
  Favorable | 13 | 15
  Neutral | 31 | 21
  Unfavorable | 3 | 7
  Extremely Unfavorable | 0 | 0

3. Secondary Outcome: Subject Preference of SC Delivery Administration of SB5 Using Questionnaire
Time Frame: at Week 6
Population: Overall number of participants analyzed means number of subjects with available assessment results
Measure: Number; unit: number of responders
Groups:
- SB5 PFS: Subject preference for the PFS at Week 6
- SB5 Pen: Subject preference for the Pen at Week 6
- No Preference: Subject who chose 'no preference' at Week 6
Arm/Group | SB5 PFS | SB5 Pen | No Preference
Number analyzed (Participants) | 46 | 46 | 46
number of responders
  Overall Preference | 14 | 26 | 6
  Category: Ease of Use | 10 | 33 | 3
  Category: Convenience | 6 | 35 | 5
  Category: Time to Administer Injection | 9 | 30 | 7
  Category: Safety | 6 | 31 | 9
  Category: Less Pain | 17 | 21 | 8

ADVERSE EVENTS:
Arm/Group | SB5 40mg
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 4/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB5 40mg (N=49)
Nasopharyngitis (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes